CLINICAL TRIAL: NCT06188572
Title: The Effect of Diabetic Peripheral Neuropathy Symptoms on Temporomandibular Joint Functionality in Patients With Type 2 Diabetes
Brief Title: The Effect of Peripheral Neuropathy Symptoms on Temporomandibular Joint Functionality
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: HRU/23.04.15
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Diabete Type 2
Keywords: diabetes mellitus; temporomandibular joint; neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes Mellitus: The study group included individuals aged 48-78 (min-max) years, diagnosed with type 2 DM in the treatment units of Harran University Training and Research Hospital.
  Interventions: Other: Michigan Neuropathy Screening Instrument; Other: Numeric Pain Scale; Other: Mandibular Function Disorder Questionnaire; Other: Fonseca Anamnestic Index; Other: Ferrans&Powers Quality of Life Index Diabetes Version
- Healthy: Age and sex homogenous healthy individuals without a diagnosis of DM were included in the control group
  Interventions: Other: Michigan Neuropathy Screening Instrument; Other: Numeric Pain Scale; Other: Mandibular Function Disorder Questionnaire; Other: Fonseca Anamnestic Index; Other: Ferrans&Powers Quality of Life Index Diabetes Version

INTERVENTIONS:
Other: Michigan Neuropathy Screening Instrument — A two-step test consisting of symptom questionnaire and physical examination was used. The symptom questionnaire includes 15 questions about the legs and feet. Physical examination includes assessment of the appearance of the feet, Achilles reflex, thumb vibration and monofilament tests.
Other: Numeric Pain Scale — In this simple method, which is frequently used to measure pain intensity in the clinic and whose validity and reliability have been demonstrated, the participant is asked to mark a number on a 10 cm scale with numbers ranging from "0" (no pain) to "10" (unbearable pain) for the pain.
Other: Mandibular Function Disorder Questionnaire — This valid and reliable scale evaluating mandibular dysfunction consists of two dimensions and 17 questions.A high total score obtained from the questionnaire indicates a high level of impairment in jaw function
Other: Fonseca Anamnestic Index — This scale, which is valid and reliable as a TMJ disorder assessment tool, includes 10 questions. The presence of TMD is accepted in those with a score of 25.
Other: Ferrans&Powers Quality of Life Index Diabetes Version — This index consists of two parts and a total of 68 items. A high score indicates a good quality of life.

SUMMARY:
The aim of this observational case-control study was to investigate the effect of diabetic peripheral neuropathy symptoms on temporomandibular joint functionality in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The number of participants planned to be included in the study was decided with the G-Power programme. While calculating the number of individuals to be included in the study, it was calculated that the sample size to obtain an effect size of 0.6 for the purpose of evaluation within the 95% confidence interval in a way to provide 80% study power at 5% Type 1 and 20% Type 2 error limits should be 74 (n=37) individuals. This study included 70 individuals (DM study group=40 individuals, control group=30 individuals).

Peripheral neuropathy symptoms of all participants were evaluated with the Michigan Neuropathy Screening Test. In the evaluation of TMJ functionality, the presence of pain, maximum pain-free mouth opening, mandibular dysfunction and dysfunction were assessed with the help of scales. Duration of diabetes mellitus was recorded and quality of life was evaluated with Ferran Powers Quality of Life Index.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type 2 DM

Exclusion Criteria:

* Having diabetic foot ulcer,
* Mini Mental Test score below 24,
* History of psychiatric illness, cancer, neurological problems, congenital anomalies, musculoskeletal problems, systemic disease, facial paralysis, surgical operation related to spine, abdomen and/or TMJ problem
* Receiving any treatment related to spine and TMJ in less than 6 months

Ages: 48 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group included individuals aged between 48-78 (min-max) years who were diagnosed with type 2 DM in the treatment units of Harran University Training and Research Hospital, while the control group included age and gender homogeneous healthy individuals without a diagnosis of DM.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Michigan Neuropathy Screening Instrument | May 2023- November 2023
  The symptom questionnaire includes 15 questions about the legs and feet. Physical examination includes assessment of the appearance of the feet, Achilles reflex, thumb vibration and monofilament tests.
  High score indicates increased neuropathy
Numeric Pain Scale | May 2023- November 2023
  The participant is asked to mark a number on a 10 cm scale, on which numbers are shown in the range of "0" (no pain) to "10" (unbearable pain) for the pain. High score indicates increased pain
Maximum pain-free mouth opening | May 2023- November 2023
  The maximum pain-free mouth opening was recorded using a 15 cm ruler
Mandibular Function Disorder Questionnaire | May 2023- November 2023
  This scale evaluating mandibular dysfunction consists of two dimensions and 17 questions.A high total score obtained from the questionnaire indicates a high level of impairment in jaw function.
Fonseca Anamnestic Index | May 2023- November 2023
  This scale includes 10 questions. The presence of TMD is accepted in those with a score of 25. High score indicates increased dysfunction.
Ferrans&Powers Quality of Life Index Diabetes Version | May 2023- November 2023
  The Quality of Life Assessment Index consists of two parts and a total of 68 items. A high score indicates a good quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Bandirma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided